CLINICAL TRIAL: NCT04129957
Title: The Prediction of Failure Rate of Dental Implants
Brief Title: Prediction of Failure of Dental Implants
Status: Completed | Type: Observational
Sponsor: Academic Centre for Dentistry in Amsterdam (Other)
Responsible Party: Principal Investigator, Naichuan Su, Principal Investigator, Academic Centre for Dentistry in Amsterdam
Other Study IDs: 2018.376
Record Dates: First submitted 2019-10-15; First posted 2019-10-17 (Actual); Last update posted 2019-10-21 (Actual); Status verified 2019-10

CONDITIONS: Implant Complication; Peri-Implantitis
Keywords: prediction; dental implants; failure; peri-implantitis
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients who underwent placement of dental implants: The study only includes one cohort. That is the patients who underwent placement of dental implants at baseline.
  Interventions: Procedure: Placement of dental implants

INTERVENTIONS:
Procedure: Placement of dental implants — All the included patients underwent the placement of at least one implant in either upper jaw, or lower jaw, or both.
  Other Names: No other intervention

SUMMARY:
The aim of the study is to identify predictors in patient profiles and implant characteristics and to develop and calibrate a prediction model for failure of implants. Patients' demographic characteristics, lifestyle habits, general health, dental health, and implant characteristics were regarded as potential predictors. The failure of implants and the follow-up time in days of implants were considered the outcome. Multivariate Cox proportional hazards regression analysis is used to find out the important risk factors for failure of dental implants and to develop the model for prediction of failure of dental implants at follow-up. The performance and clinical values of the model is determined.

DETAILED DESCRIPTION:
During the past decades, dental implant therapy has developed into a successful treatment option for patients confronted with both partial and complete edentulism. Based on the literature, the survival rate of dental implants, which is defined that the dental implants are still in the mouth after insertion, is around 95% in the 5-year follow-up and around 90% in the 10-year follow-up. The success rate of dental implants, which is defined as dental implants in function, with good hard and soft tissue physiology and user satisfaction ranges from 85.2% to 88.7% in the follow-up of up to 20 years. This indicates that both the success rate and survival rate of dental implants is high. However, both survival rates and success rates vary across patients with different profiles. The expense of dental implant treatment is high and implant placement is a surgical procedure which is invasive and thus risky for the patients' health. Once the failure of dental implants occurs, it may cause some severe negative consequences for patients. For example, the failure will cause a financial loss for patients and a possible shock concerning both mental and physical aspects. To reduce these risks it is important and necessary for clinicians to be able to predict the risk of the failure of dental implants of individual patients before they undergo dental implant treatment.

Aim:

The aim of the project is to find out the possible risk factors for failure of dental implants and to develop a prediction model for the failure of dental implants at follow-up as a tool for clinicians to establish patients individual risk profile.

Methods:

The study is a retrospective design. The clinical data of the adult patients who were referred to the Department of Oral Implantology and Prosthetic Dentistry, Academic Centre for Dentistry Amsterdam (ACTA) for placement of dental implants from September 2009 to September 2013 are collected retrospectively from the clinical data management system of ACTA in the study.

The potential predictors include five domains: patients' demographic characteristics, lifestyle habits, general health, dental health, and implant characteristics. These predictors are pre-screened by international experts in dental implantology based their clinical knowledge and experience.

The outcomes included the follow-up time of implants and whether the failure of the implants was observed at the follow-up. The follow-up time is defined as the difference in time between implant placement and implant failure, or the date of the last follow-up time point if the dental implant is in an acceptable state. The failure of implants is defined as the presence of peri-implantitis, presence of mobility of implants, or removal of the implants for any reasons, for instance, unacceptable performance in aspects of function, tissue physiology, esthetics, and patients' satisfaction after placement of suprastructure.

The Multivariate Cox proportional hazards regression analysis will be used to find out the important risk factors and to develop the model. The performance of the model, in aspects of calibration and discrimination, is assessed. The clinical added values of the model is assessed. Then, the model is transformed into a score chart and a line chart, which is easy-to-use to the clinicians for the prediction.

ELIGIBILITY:
Inclusion Criteria:

* patients were over 18 years old at baseline;
* patients underwent the placement of at least one implant;
* patients were followed up for the implants at least one time after placement of implants;
* patients provided their informed consent.

Exclusion Criteria:

* patients were <18 years old at baseline;
* patients were not followed up;
* patients did not provide the informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The included patients were those who were referred to the Department of Oral Implantology and Prosthetic Dentistry, ACTA for placement of implant(s).
Sampling Method: Probability Sample
Enrollment: 337 (Actual)
Dates: Start 2018-12-10 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-08-15 (Actual)

PRIMARY OUTCOMES:
Failure of dental implants | up to 5 years follow-up
  The failure of implants was defined as the presence of peri-implantitis, presence of mobility of implants, or removal of the implants for any reasons, for instance, unacceptable performance in aspects of function, tissue physiology, esthetics, and patients' satisfaction after placement of suprastructure.
Follow-up time | up to 5 years follow-up
  The follow-up time is defined as the difference in time between implant placement and implant failure, or the date of the last follow-up time point if the dental implant is in an acceptable state.

CONTACTS AND LOCATIONS:
Overall Officials: Geert van der Heijden, Prof. dr., Study Chair — Academic Centre for Dentistry Amsterdam
Locations (1):
- Academic Centre for Dentistry in Amsterdam, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
The participants' clinical data and data on demographic characteristics are possible to be shared. But those data can be only used for research purpose.
Supporting Information: Study Protocol, SAP
Time Frame: Starting 6 months after the publication. The data will be available for 15 years after the end of the study.
Access Criteria: The data can be shared upon researchers' request via email (n.su@acta.nl). Naichuan Su will review the requests. The researchers need to share their protocols and guarantee that the data is only used for research purpose.

REFERENCES:
- [Background] Pjetursson BE, Thoma D, Jung R, Zwahlen M, Zembic A. A systematic review of the survival and complication rates of implant-supported fixed dental prostheses (FDPs) after a mean observation period of at least 5 years. Clin Oral Implants Res. 2012 Oct;23 Suppl 6:22-38. doi: 10.1111/j.1600-0501.2012.02546.x. PMID 23062125
- [Background] Pjetursson BE, Asgeirsson AG, Zwahlen M, Sailer I. Improvements in implant dentistry over the last decade: comparison of survival and complication rates in older and newer publications. Int J Oral Maxillofac Implants. 2014;29 Suppl:308-24. doi: 10.11607/jomi.2014suppl.g5.2. PMID 24660206
- [Background] Jung RE, Zembic A, Pjetursson BE, Zwahlen M, Thoma DS. Systematic review of the survival rate and the incidence of biological, technical, and aesthetic complications of single crowns on implants reported in longitudinal studies with a mean follow-up of 5 years. Clin Oral Implants Res. 2012 Oct;23 Suppl 6:2-21. doi: 10.1111/j.1600-0501.2012.02547.x. PMID 23062124
- [Background] Krebs M, Schmenger K, Neumann K, Weigl P, Moser W, Nentwig GH. Long-term evaluation of ANKYLOS(R) dental implants, part i: 20-year life table analysis of a longitudinal study of more than 12,500 implants. Clin Implant Dent Relat Res. 2015 Jan;17 Suppl 1:e275-86. doi: 10.1111/cid.12154. Epub 2013 Sep 17. PMID 24103113
- [Background] Lekholm U, Grondahl K, Jemt T. Outcome of oral implant treatment in partially edentulous jaws followed 20 years in clinical function. Clin Implant Dent Relat Res. 2006;8(4):178-86. doi: 10.1111/j.1708-8208.2006.00019.x. PMID 17100743
- [Background] Ostman PO, Hellman M, Sennerby L. Ten years later. Results from a prospective single-centre clinical study on 121 oxidized (TiUnite) Branemark implants in 46 patients. Clin Implant Dent Relat Res. 2012 Dec;14(6):852-60. doi: 10.1111/j.1708-8208.2012.00453.x. Epub 2012 May 29. PMID 22642261

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-09-21): https://cdn.clinicaltrials.gov/large-docs/57/NCT04129957/Prot_SAP_ICF_000.pdf